CLINICAL TRIAL: NCT02654262
Title: Obesity and Bone Development in Young Girls
Brief Title: Soft Tissue and Bone Development in Young Girls
Acronym: STAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: HD74565
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Bone Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
Obesity during adolescence, a critical time for bone development, may impair mineral accrual and reduce bone strength, leading to greater fracture risk during adolescence and later in life. This study seeks to determine the effect of obesity and accompanying metabolic changes (insulin resistance and inflammation) on bone mineral accrual and related changes in structure and strength in young girls. The information is critical to developing effective prevention strategies to counter the linked risks of obesity and osteoporosis, both major public health concerns.

DETAILED DESCRIPTION:
The pediatric obesity epidemic continues unabated. Its cardio-metabolic complications are undisputed, including inflammation, insulin resistance (IR), glucose intolerance and greater prevalence of type 2 diabetes (T2D) in youth. We contend an equally serious consequence of these obesity co-morbidities is their detrimental effects on bone development during adolescence, a critical time for mineral accrual and architectural modeling that underlies bone strength and fracture risk. This proposition has received little attention and the sparse results are mixed, with reports of augmented and impaired mineralization. In contrast, animal data demonstrates reduced mineral accrual and compromised architecture with insulin resistance and chronic inflammation. The conflicting results in youth are likely due to mixed samples and analyses that commingle obese youth with metabolic complications with so called metabolically healthy obese youth and the use of technology (i.e., dual energy x-ray absorptiometry, DXA) to measure bone outcomes that is confounded by the very changes that investigators seek to detect. We posit that the positive mechanical effect of excess adiposity on bone is countered by chronic low-grade inflammation and IR so that obese youth with these metabolic complications suffer impaired bone development whereas obesity in otherwise metabolically healthy youth augments development. A thorough understanding of the effects of adiposity and its co-morbidities on bone development is crucial to the development of efficacious interventions aimed at maximal mineral accrual and bone modeling. Thus, we propose primary aims designed to clarify the effects of obesity, insulin resistance and inflammation on bone around the time of peak height velocity. Adipose tissue (AT) distribution undoubtedly matters, especially abdominal visceral AT and skeletal muscle fat content, both strongly related to insulin resistance. Failure to characterize fat distribution is another important limitation of past studies. Consequently we will assess the effect of visceral AT and skeletal muscle fat along with whole body fatness and propose secondary aims designed to develop safe, cost effective methods that we and others can use for estimating AT distribution, a critical component of risk that has rarely been studied in youth relative to bone development.

Primary Aims:

1. Assess the associations of total and regional adiposity (visceral AT and leg muscle fat content), insulin resistance, and inflammation with bone mass, density, structure and strength in normal weight, overweight, and obese pre-menarcheal girls
2. Assess the effects of total and regional adiposity, insulin resistance, and inflammation on bone development (i.e., 2 year changes in bone parameters) in normal weight and obese pre-menarcheal girls.

ELIGIBILITY:
Inclusion Criteria:

* healthy, female, aged 9-12 years

Exclusion Criteria:

* diagnosis of diabetes
* taking medications that alter body composition and bone mineral accrual
* physical disability that limits physical activity
* learning disability that would limit completion of questionnaires

Ages: 9 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Girls across obese (n=150; BMI ≥95th age and gender-specific percentile), overweight (n=150; BMI> 85th percentile and <95th percentile), and normal weight (n=150; BMI< 85th percentile) categories.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Bone development | 2 years
  Baseline cross-sectional (N=450) and longitudinal changes over 2 years (N=150) in bone mass, density, structure and strength, measured by peripheral quantitative computed tomography (pQCT) and dual-energy X-ray absorptiometry (DXA), as they relate to body composition by DXA and blood biomarkers of insulin resistance and inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Going, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Nutritional Sciences Department, Tucson, Arizona, United States

REFERENCES:
- [Derived] Hetherington-Rauth M, Bea JW, Lee VR, Blew RM, Funk J, Lohman TG, Going SB. Comparison of direct measures of adiposity with indirect measures for assessing cardiometabolic risk factors in preadolescent girls. Nutr J. 2017 Feb 23;16(1):15. doi: 10.1186/s12937-017-0236-7. PMID 28231807